CLINICAL TRIAL: NCT02131220
Title: A Randomized, Parallel-controlled, Multi-center Study of the Effects of Intracoronary Recombinant HUman Prourokinase or TIrofiban on the Coronary Flow During Primary PCI for the Acute Myocardial InfartiON
Brief Title: Effects of Intracoronary Prourokinase on the Coronary Flow During Primary Percutaneous Coronary Intervention for Acute Myocardial Infarction
Acronym: ERUPTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ge Junbo, Director, Dept. of Cardiology, Shanghai Institute of Cardiovascular Diseases, Zhongshan Hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Zhongshan 2012-134
Record Dates: First submitted 2014-05-03; First posted 2014-05-06 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Myocardial Infarction; Percutaneous Coronary Intervention; Thrombolytic Therapy
Keywords: No-Reflow Phenomenon
MeSH Terms: conditions — Myocardial Infarction; No-Reflow Phenomenon | interventions — saruplase; Injections; Tirofiban; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Prourokinase (Experimental): Intracoronary bolus infusion of 20mg prourokinase using selective catheter
  Interventions: Drug: Prourokinase
- Tirofiban (Active Comparator): Intracoronary tirofiban bolus infusion using selective catheter (10ug/kg)
  Interventions: Drug: Tirofiban
- Normal saline (Placebo Comparator): Intracoronary saline bolus infusion using selective catheter (20ml)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Prourokinase — 20mg intracoronary bolus infusion using selective catheter during PCI
  Other Names: Reocmbinant Human Prourokinase for Injection; TIANJIN TASLY PHARMACEUTICAL CO.,LTD
  Arms: Prourokinase
Drug: Tirofiban — 10ug/kg intracoronary bolus infusion using selective catheter during PCI
  Other Names: Grand Pharmr (China) Co. Ltd
  Arms: Tirofiban
Drug: normal saline — intracoronary bolus infusion using selective catheter during PCI
  Arms: Normal saline

SUMMARY:
The purpose of this study is to determine whether intracoronary selective thrombolysis are more effective than tirofiban on the coronary flow during primary percutaneous coronary intervention for the acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* ST-segment elevation AMI within 12 hours of symptom onset

Exclusion Criteria:

* Contraindications to thrombolysis or PCI
* Patients administered a fibrinolytic agent before PCI
* Patients enrolled in clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Coronary flow using corrected Thrombolysis In Myocardial Infarction Frame Count (cTFC) | At the end of Percutaneous Coronary Intervention procedure

SECONDARY OUTCOMES:
ST segment resolution in ECG | 3 hours post PCI procedure
peak troponin T level | in the 7 days post PCI procedure
plasma N terminal-proBNP levels | 1 and 30 days post PCI procedure
infarction area confirmed by SPECT | 30 days post PCI
incidence of major adverse cardiac events (MACE) defined as the composite of death, myocardial infarction and target vessel revascularization | 30 days post PCI

OTHER OUTCOMES:
TIMI defined total major bleeding | 30 days post PCI

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, M.D., Principal Investigator — Department of Cardiology, Zhongshan Hospital, Fudan University
Locations (1):
- Department of Cardiology, Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China